CLINICAL TRIAL: NCT03505398
Title: Study of Visual-spatial Attention by Oculomotor Recording (Eye Tracking) as a Function of Central or Peripheral Visual Impairment
Brief Title: Study of Visual-spatial Attention by Eye Tracking as a Function of Central or Peripheral Visual Impairment
Acronym: BEHAVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Despite an extension of the planned duration of inclusion and an enrolled patient number inferior than planned, coordinating investigator considered that it was more reasonable to stop inclusions in order to analyze the data already available
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC17_0134; 2017-A00977-46 (Other: ANSM)
Record Dates: First submitted 2018-03-27; First posted 2018-04-23 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Central or Peripheral Visual Impairment
MeSH Terms: interventions — Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- central vision disorder (Experimental)
  Interventions: Procedure: microperimetry; Procedure: visual acuity; Procedure: automated visual field; Procedure: eye movements recording
- peripheral vision disorder (Experimental)
  Interventions: Procedure: microperimetry; Procedure: visual acuity; Procedure: automated visual field; Procedure: eye movements recording
- control (Other)
  Interventions: Procedure: microperimetry; Procedure: visual acuity; Procedure: automated visual field; Procedure: eye movements recording

INTERVENTIONS:
Procedure: microperimetry — define the retinal fixation point and the differential sensitivity threshold of the retina.
Procedure: visual acuity — using ETDRS scales
Procedure: automated visual field — recording visual attention based on central or peripheral visual information
Procedure: eye movements recording — recording of explicit visual attention based on central or peripheral visual information

SUMMARY:
The objective of this pilot work is to determine the role of central and peripheral visions in explicit attention processes (saccade planning) in the case of visual impairment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years;
* Patient with a central visual deficit (central scotoma on the visual field: DMLA, cones dystrophy ...) or peripheral (annular scotoma: chronic glaucoma, retinitis pigmentosa ...) or without visual deficit (corrected visual acuity and visual field)
* Patient agreeing to participate in the study and signing informed consent
* Patient affiliated to social security

Exclusion Criteria:

* Pregnant woman
* Patient with known epilepsy
* Major under judicial safeguard, or deprived of liberty
* Major under guardianship or curatorship or admitted to a health or social institution for purposes other than research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Measurement of visual acuity (central versus peripheral) | Day 0
Microperimetry recording (central versus peripheral) | Day 0
recording of automated visual field (central versus peripheral) | Day 0
recording of eye movements (central versus peripheral) | Day 0

SECONDARY OUTCOMES:
Measurement of visual acuity (patient versus control) | Day 0
Microperimetry recording (patient versus control) | Day 0
recording of automated visual field (patient versus control) | Day 0
recording of eye movements (patient versus control) | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France